CLINICAL TRIAL: NCT01242982
Title: Prospective Randomised Study of Subcapital and Shaft Fractures of the 5. Metacarpal. Comparison Conservative Treatment and Operation
Brief Title: Subcapital and Shaft Fractures of the 5. Metacarpal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: problems to include patients, patients not showing up at check-up
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOSL-2010
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Fracture
Keywords: 5. metacarpal fracture/fractures; subcapital; shaft; closed
MeSH Terms: conditions — Fractures, Bone | interventions — Calcium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operation (Experimental): Closed reduction and operated for fixation with 2 antegrade intramedullary Kirschner wires.
  Interventions: Procedure: Closed reduction and fixation with 2 pins
- Conservative treatment (Active Comparator): Treated conservatively with reduction and then Plaster of Paris.
  Interventions: Procedure: Reduction and Plaster of Paris

INTERVENTIONS:
Procedure: Closed reduction and fixation with 2 pins — Closed reduction and fixation with 2 antegrade intramedullary Kirschner wires. Cast for 2 weeks. Control after 2 and 5 weeks. Thereafter a control after 3,6 and 12 months
  Arms: Operation
Procedure: Reduction and Plaster of Paris — Closed reduction in local anesthesia and a Plaster of Paris for max. 3 weeks. Control after 1 and 3 weeks, thereafter control after 3,6 and 12 months
  Arms: Conservative treatment

SUMMARY:
The purpose of this study is to find out the best treatment for subcapital and shaft fractures of the 5. metacarpal.

It is a prospective randomized multicenter study. Comparing only fractures dislocated more than 30 degrees.

One group will be operated with intramedullary pins and one group will be treated conservatively with reduction and then Plaster of Paris for 3 weeks.

All patients will be followed up after 3, 6 and 12 months.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* voluntarily, only isolated subcapital og shaft fracture of the 5. metacarpal,operated/reduction within 10 days of injury,not intoxicated,degree of fracture dislocation minimum 30 degrees measured on the X-ray.

Exclusion Criteria:

* open fractures, fractures of the head of 5. metacarpal/intraarticular fractures, patients who wants to be followed up at Hospitals outside the study area, earlier injury of the hand that might have influence on function.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Clinical outcome comparing conservative and operative treatment of subcapital and shaft fractures of the 5. metacarpal | 2 -3 years
  The goal is 200 patients with shaft and subcapital fractures of the 5.metacarpal. In each group the goal is 100 patients there 50 patients will be operated (2 intramedullary pins) and 50 patients undergo conservative treatment. The follow up is 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Rossvoll, dr. med., Study Director — St. Olavs Hospital, orthopedic department
Locations (5):
- Norway (5):
  - Ålesund sjukehus, Helse Sunmøre, Ålesund, Møre og Romsdal
  - Kristiansund sykehus, Helse Nord Møre og Romsdal, Kristiansund-N, Møre og Romsdal
  - Molde sykehus, Helse Nordmøre og Romsdal, Molde, Møre og Romsdal
  - Sykehuset Namsos, Helse Nord-Trøndelag, Namsos, Nord -Trøndelag
  - Sykehuset i Vestfold-Tønsberg, Tønsberg